CLINICAL TRIAL: NCT01635192
Title: Effects of Probiotic VSL#3 on Expression of Small Intestinal Mucosal Renin-angiotensin System and Glucose Absorption in Man - a Doubleblind, Randomized Parallel Arm Placebo Controlled Exploratory Study in Healthy Volunteers
Brief Title: Effects of Probiotic VSL#3 on Expression of Small Intestinal Renin-angiotensin System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ProGlucose-1
Record Dates: First submitted 2012-06-28; First posted 2012-07-09 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2014-05

CONDITIONS: the Local Renin-angiotensin System (RAS) in Small Intestinal Mucosa in Man
Keywords: renin; angiotensin; probiotic; glucose absorption; intestinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Active Comparator)
  Interventions: Biological: VSL#3
- Inactive treatment (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VSL#3 — The probiotic product VSL#3® comes in a powder (sachet) that is to be dissolved in half a glass of cold water before ingestion. Two sachets are ingested once daily over 2 weeks.
  Each dose (sachet) contains 450 billion live (lyophilized) lactic acid bacteria (in defined ratios of the following strains: Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, Lactobacillus bulgaricus, Streptococcus thermophilus) and are delivered in a base of maltose and silicon dioxide.
  Arms: VSL#3
Biological: Placebo — Two placebo sachets containing maltose and silicon dioxide are given once daily over 2 weeks.
  Arms: Inactive treatment

SUMMARY:
Probiotics have become very popular and are by WHO defined as "Live microorganisms which when administered in adequate amounts confer a health benefit on the host". For example, probiotics have been shown to contribute to improvements of abdominal discomfort and intestinal inflammation. The main hypothesis behind the present study is that probiotics influences mucosal regulatory systems, particularly the actions of the hormone Angiotensin II locally in the intestinal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers of both sexes
* between 18 and 65 years of age.
* BMI between 18-25 kg/m2

Exclusion Criteria:

* Any drug abuse
* Use of prescription medication within the previous 14 days (with the exception of contraceptives)
* Pregnant or breast feeding woman or woman of childbearing potential not using adequate birth control (e.g. IUD, barrier method, oral contraceptive, abstinence)
* In the investigator's judgement, clinically significant abnormalities at the screening examination or in the laboratory test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The change in mucosal expression of components of renin-angiotensin (particularly ACE1, AT1-receptor, AT2-receptor) | Change from baseline in protein expressions after 2 weeks of treatment.
  Mucosal biopsies from jejunum are sampled via endoscopy immediately before (baseline) and at the end of the 2 weeks treatment period. Protein expressions are assessed by western blotting and the subject acts as its own control.

SECONDARY OUTCOMES:
Changes in epithelial permeability and glucose absorption capacity in vitro | Change from baseline at 2 weeks after start of treatment.
  Mucosal biopsies are mounted in modified Ussing chambers. Permeability and glucose-absorption are assessed.
Change in intestinal glucose absorption capacity in-vivo | Change from baseline at 2 weeks after start of treatment.
  Glucose (75g) with an non-metabolisable analogue (3-O-methyl-glucose; 2g) is instilled into the duodenum via a nasogastroduodenal tube (corresponding to an oral glucose tolerance test). Plasma glucose, 3OMG and insulin are assessed in 15 min periods over 2h.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Dept of Gastrosurgical R&E, Sahlgrenska Universityhospital, Gothenburg, Sweden